CLINICAL TRIAL: NCT05847387
Title: Preoperative Surgeon Evaluation of Corneal Endothelial Status: the Viability Control of Human Endothelial Cells Before Keratoplasty (V-CHECK) Study
Brief Title: The Viability Control of Human Endothelial Cells Before Keratoplasty (V-CHECK) Study
Acronym: V-CHECK
Status: Recruiting | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Vito Romano, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: VC1
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Corneal Transplant Failure; Corneal Endothelial Cell Loss
Keywords: Keratoplasty; Corneal endothelium; Eye Banking
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Keratoplasty group: Patients undergoing keratoplasty and their respective donor tissue
  Interventions: Diagnostic Test: V-Check

INTERVENTIONS:
Diagnostic Test: V-Check — Preoperative analysis of endothelial tissue staining with vital dye (Trypan Blue 0.05%) and image analysis to identify the percentage of Trypan Blue Positive Areas, corresponding to dead endothelial cells and/or denuded areas of endothelium, in tissues destined to keratoplasty

SUMMARY:
The purpose of this international cohort study is to validate a new method for preoperative assessment of endothelial viability in donor corneal tissues for transplantation, and to correlate endothelial health as assessed by the surgical team to functional and structural long-term outcomes in the cohort of patients receiving them.

DETAILED DESCRIPTION:
The corneal endothelium is responsible for preserving corneal transparency by maintaining a dynamic equilibrium of corneal stromal hydration. Corneal Endothelial Cells (CECs) health is approximated by evaluating the Endothelial Cell Density (ECD) of corneal tissues though specular biomicroscopy. ECD is a key determinant of long-term tissue survival after corneal transplantation, as corneal graft function is directly dependent on the number of viable CECs. However, ECD represents only an estimation of total corneal endothelial health and is a suboptimal proxy for future endothelial failure.

In the current chain of supply of donor corneal tissues, no independent evaluation of endothelial cell viability by the surgical team tasked with transplanting the donor corneal tissue is anticipated. The investigators have previously shown a poor correlation between ECD declared by the eye bank providing the tissue and tissue quality as assessed independently by a cornea surgeon performing the transplantation (unpublished data).

In this study, the investigators describe a simple method to independently evaluate the overall endothelial viability of donor corneal tissue which can be adopted both by eye banks before shipment and by the corneal surgeons before transplantation in the operating theatre. This method uses basic image analysis to assess the extent of endothelial cell death and/or denuded endothelial areas with the use of Trypan Blue, a vital dye commonly employed during corneal transplantation. Endothelial cell loss is visualized and quantified as Trypan Blue Positive Areas (TBPA).

The primary objective of this study is to quantify the extent of TBPA in the operating theatre before corneal transplantation and correlate it to overall donor mortality declared by the eye bank. Secondary objectives include the assessment of the correlation of TBPA with declared ECD and CECs mortality, on folds, as well as the longitudinal analysis of endothelial cell loss as a function of time from surgery and initial TBPA over a follow-up of 12 months, final ECD, incidence of graft failure, and risk of graft failure attributable to preoperative TBPA.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old
* Planned corneal transplantation: perforating keratoplasty (PK), Descemet stripping automated endothelial keratoplasty (DSAEK), ultra-thin DSAEK (UT-DSAEK) or Descemet membrane endothelial keratoplasty (DMEK)
* Indication for corneal transplantation (low-moderate risk of rejection): keratoconus, Fuchs endothelial dystrophy
* Ability to provide written informed consent.

Exclusion Criteria:

* Prior corneal transplantation
* Planned preloaded DSAEK or preloaded DMEK
* Planned keratoplasty not involving corneal endothelium transplantation (i.e., superficial/deep anterior lamellar keratoplasty)
* Evidence of concurrent microbial keratitis
* Evidence of non-infectious or autoimmune keratitis
* Impending or frank corneal perforation
* Uncontrolled, elevated intraocular pressure (IOP)- Previous glaucoma surgery
* Acute or chronic inflammatory/infectious anterior segment uveitis
* Presence of an anterior chamber intraocular lens (IOL) for phakic or aphakic purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing keratoplasty at participating referral cornea clinics
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Trypan Blue Positive Areas (TBPA) percentage and Donor mortality | Preoperative
  The comparison of the endothelial mortality of included donor corneas measured preoperatively (TBPA) and the overall endothelial mortality as declared by the eye bank providing the tissue

SECONDARY OUTCOMES:
Correlation of TBPA to declared endothelial cell density (dECD) | Preoperative
  Spearman's rank correlation coefficient of TBPA and declared Endothelial Cell Density (dECD) as provided by the Eye Bank supplying the tissue
Correlation of TBPA to declared endothelial mortality on corneal folds | Preoperative
  Spearman's rank correlation coefficient of TBPA and declared Endothelial Cell mortality on corneal folds as provided by the Eye Bank supplying the tissue
Final ECD | 1 year after enrollment
  Final ECD of transplanted corneas at 12 months
Rate of endothelial cell loss | 1 year after enrollment
  Rate of change of ECD over the course of the entire follow-up
Incidence of endothelial graft failure | 1 year after enrollment
  The occurrence of clinically definite corneal edema and/or need for endothelial keratoplasty due to endothelial failure
Relative risk of endothelial graft failure associated with TBPA | Preoperative
  Calculation through a proportional hazard model of the relative risk of endothelial graft failure attributable to preoperatively measured TBPA

CONTACTS AND LOCATIONS:
Overall Officials: Vito Romano, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Locations (12):
- Antwerp University Hospital, Edegem, Belgium
- Germany (2):
  - Department of Ophthalmology, University of Cologne, Cologne
  - Münster University Hospital, Münster
- Italy (6):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia, BS
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Department of Medical and Surgical Sciences, University Magna Græcia, Catanzaro
  - Department of Experimental Medicine, Tor Vergata School of Medicine and Surgery, Roma
  - Fondazione Banca degli Occhi del Veneto, Venice
  - San Bortolo Hospital, Vicenza
- Maastricht University Medical Center, Maastricht, Netherlands
- Hospital Regional Universitario de Málaga, Málaga, Spain
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD with appropriated anonymization of sensible data will be stored to a dedicated repository after completion of the study
Supporting Information: Study Protocol
Time Frame: After completion of study
Access Criteria: Upon approval of individual sharing request

REFERENCES:
- [Derived] Airaldi M, Zheng Y, Aiello F, Bachmann B, Baydoun L, Ni Dhubhghaill S, Dickman MM, Kaye SB, Fontana L, Gadhvi KA, Moramarco A, Rodriguez Calvo de Mora M, Rocha de Lossada C, Scorcia V, Viola P, Calza S, Levis HJ, Parekh M, Ruzza A, Ferrari S, Ponzin D, Semeraro F, Romano V. Preoperative surgeon evaluation of corneal endothelial status: the Viability Control of Human Endothelial Cells before Keratoplasty (V-CHECK) study protocol. BMJ Open Ophthalmol. 2023 Sep;8(1):e001361. doi: 10.1136/bmjophth-2023-001361. PMID 37730252